CLINICAL TRIAL: NCT07364253
Title: Clinical Evaluation Of The Effects Of Propolis Gargle On Wound Healing After Impacted Third Molar Surgery
Brief Title: 'Propolis Versus Chlorhexidine Gluconate on Wound Healing After Third Molar Surgery: a Randomized Controlled Trial'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Zeynep Bayramoglu, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/3-4
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Third Molar Surgery; Post Operative Analgesia
Keywords: third molar surgery; propolis gargle; chlorhexidine gluconate
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis gargle (Active Comparator): Patients were randomly allocated into two groups: one group used 0.12% chlorhexidine gluconate gargle, while the other used a 3% propolis-containing gargle. Gargles were applied twice daily for one minute from postoperative day 2 to day 7. Pain was evaluated using the visual analog scale (VAS), while edema, maximum mouth opening, wound healing, and postoperative complications were assessed preoperatively and on postoperative days 2 and 7.
  Interventions: Procedure: Third molar Surgery with propolis gargle
- Chlorhexidine Gluconate gargle (Active Comparator): Patients were randomly allocated into two groups: one group used 0.12% chlorhexidine gluconate gargle, while the other used a 3% propolis-containing gargle. Gargles were applied twice daily for one minute from postoperative day 2 to day 7. Pain was evaluated using the visual analog scale (VAS), while edema, maximum mouth opening, wound healing, and postoperative complications were assessed preoperatively and on postoperative days 2 and 7.
  Interventions: Procedure: Third molar surgery with chlorhexidine gluconate

INTERVENTIONS:
Procedure: Third molar Surgery with propolis gargle — The patients were anesthetized with inferior alveolar, lingual, and buccal nerve blocks using 4 ml of articaine with 1:100,000 epinephrine (Ultracaine D-S Fort, Aventis). The tooth could be observed by elevating a full-thickness triangular mucoperiosteal flap. The tooth was extracted following an osteotomy using a bur. The tooth was sectioned and extracted, if required. Curettage was conducted in the presence of a residual dental follicle. The wound was sutured with silk thread. All procedures were conducted by the same physician. Postoperatively, antibiotics (amoxicillin combined with clavulanic acid, 2 g daily for 5 days) and analgesics (paracetamol 1 g, up to 4 times daily for 3 days) were recommended. The group was administered a 3% propolis gargle (formulated in an ethanol solution, twice daily for 1 minute, prepared in the Departments of Pharmacology.
  Arms: Propolis gargle
Procedure: Third molar surgery with chlorhexidine gluconate — The patients were anesthetized with inferior alveolar, lingual, and buccal nerve blocks using 4 ml of articaine with 1:100,000 epinephrine (Ultracaine D-S Fort, Aventis). The tooth could be observed by elevating a full-thickness triangular mucoperiosteal flap. The tooth was extracted following an osteotomy using a bur. The tooth was sectioned and extracted, if required. Curettage was conducted in the presence of a residual dental follicle. The wound was sutured with silk thread. All procedures were conducted by the same physician. Postoperatively, antibiotics (amoxicillin combined with clavulanic acid, 2 g daily for 5 days) and analgesics (paracetamol 1 g, up to 4 times daily for 3 days) were recommended. The group was administered chlorhexidine gluconate (0.12%) gargle, twice daily for 1 minute.
  Arms: Chlorhexidine Gluconate gargle

SUMMARY:
The goal of this study is to examine the effects of propolis gargle on wound healing following third molar surgery and to compare it with chlorhexidine gluconate. The main question it aims to answer is:

Is propolis-containing gargle safe and effective alternative to chlorhexidine gluconate following impacted third molar surgery? Does propolis demonstrate comparable outcomes in pain control and mouth opening ?

DETAILED DESCRIPTION:
This prospective, randomized clinical study included 52 healthy patients (ASA I) who underwent impacted mandibular third molar surgery. Patients were randomly allocated into two groups: one group used 0.12% chlorhexidine gluconate gargle, while the other used a 3% propolis-containing gargle. Gargles were applied twice daily for one minute from postoperative day 2 to day 7. Pain was evaluated using the visual analog scale (VAS), while edema, maximum mouth opening, wound healing, and postoperative complications were assessed preoperatively and on postoperative days 2 and 7. Statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of the impacted teeth were classified as Class II level B mesioangular position
* Patients from a socioeconomic level who can actively use postoperative gargles

Exclusion Criteria:

* Individuals with third molars exhibiting acute infection
* smokers
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Edema | Before surgery to after surgery seventh day
  Edema (assessed by measuring the distances between the tragus and lip corner, as well as the outer corner of the eye and mandibular corner, with measurements taken twice using a paper ruler and averaged), It was measured before surgery, after surgery second and seventh days.
Pain after surgery | After surgery, post- op second and seventh day
  Patient records were collected on the second and seventh days post-operation. The evaluated parameters included pain (measured using the VAS scale). Visual analog scale is used to measure pain intensity. It consists of a straight line usually 10 cm. 0: no pain, 10: worst pain imaginable. The patient marks the point that best represents their pain.

SECONDARY OUTCOMES:
Maximum mouth opening | Before surgery to post surgery seventh day
  Maximum mouth opening (the distance between the lower and upper incisors) were measured before surgery and after surgery second and seventh day.
Wound aperture | From surgery to seventh day after surgery
  Wound aperture after surgery was examined for two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Faculty of Dentistry, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No